CLINICAL TRIAL: NCT04060537
Title: A Retrospective Translational Study to Identify Novel Biomarkers of Response to Systemic Treatments in Renal Cell Cancer
Brief Title: Identification of Novel Biomarkers of Response to Systemic Treatments in Renal Cell Cancer
Acronym: ARTIST_RCC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: CCTU- Cancer Theme (Other)
Responsible Party: Sponsor-Investigator, CCTU- Cancer Theme, Dr. Sarah J. Welsh, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Other Study IDs: ARTIST RCC
Record Dates: First submitted 2019-08-13; First posted 2019-08-19 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Carcinoma, Renal Cell
Keywords: Cancer; Renal; Tyrosine Kinase Inhibitors; Systemic Treatments; Biomarkers
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Renal Cell Carcinoma tumour specimen (tissue block or slides), kidney tissue specimen (tissue block or slides), previously obtained with consent under NeoSUN study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Research: Patients with Renal Cell Carcinoma who have had previous systemic treatment, with adequate tissue samples and radiological data
  Interventions: Other: Laboratory analysis of samples; Other: Application of machine learning

INTERVENTIONS:
Other: Laboratory analysis of samples — RNA sequencing, immunohistochemistry, immunofluorescence, and cytometry of tumour tissues
Other: Application of machine learning — Using machine learning to interrogate data generated from analysis of Renal Cell Cancer tumours using RNA sequencing, immunohistochemistry, immunofluorescence, cytometry, and MRI imaging of tumours.

SUMMARY:
This research study aims to investigate changes inside kidney cancers (also known as Renal Cell Carcinoma or RCC), and in normal kidney surrounding the tumour, when patients are treated with systemic therapy.

Samples, radiological images and data from a previous trial (NeoSUN) will be analysed and/or reanalysed, in accordance with the consent of NeoSUN participants.

DETAILED DESCRIPTION:
This research study aims to investigate changes inside kidney cancers, and in normal kidney surrounding the tumour, when patients are treated with systemic therapy. Systemic treatment is widely used as routine treatment for patients who have kidney cancer that has spread to other organs. It is also used sometimes before surgery to try to shrink kidney cancers to make surgery easier and less risky. Recent research has shown that kidney cancers consist of many different cells in addition to the cancer cells (including immune, structural and blood vessel cells). However, doctors know very little about what changes systemic therapy causes to cells other than cancer cells.

Researchers now think that these other cells may influence how the tumour cells behave during cancer treatment and how well the cancer responds to treatment.

The NeoSUN clinical trial was run at Cambridge University Hospitals between 2006 and 2015.18 patients were treated with a TKI called sunitinib for 12 days before they had their kidney surgically removed. MRI and CT scans were performed before and after the treatment. Samples of tumour and normal kidney were also taken before and after treatment. All patients consented to use of their tissue and data for future research projects. The investigators would like to analyse the effects that sunitinib had on the tumour and other cells using techniques called immunohistochemistry, immunofluorescence, and CyTOF. These mark the different cells so they can easily be identified and the effects on each one analysed. The investigators would also like to re-analyse the scans performed and use artificial intelligence (AI) to see try to detect new trends. The information may help to guide which drugs might be best used in future to treat kidney cancer more effectively whilst keeping side effects low.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older
2. Diagnosis of renal cell cancer (any stage).
3. Patient received systemic treatment for their renal cancer at Cambridge University Hospitals NHS Foundation Trust.
4. Patients must have consent in place, for the use of tissue and imaging to be used for the purposes of clinical research;

   * Use of tissue not required for their diagnosis or treatment to be stored and used for the purposes of clinical research, which may include genetic research.
   * Use of relevant sections of their medical records, or by relevant regulatory authorities, where my tissue is being used for research, giving permission for those individuals to have access to their medical records.
5. Participants must also meet at least one of the following criteria to be eligible:

   1. For tissue analysis: Patient must have tumour tissue and/or normal adjacent kidney stored (either as formalinfixed paraffin-embedded tissue, or as 'fresh frozen' tissue).
   2. For imaging analysis: Patient must have had at least 1 scan (either CT or MRI) within 28 days of starting treatment with systemic treatment for their cancer.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with renal cell cancer who have given prior consent under NeoSUN for their samples and data to be used, and who have adequate samples and data available.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Biological identification of biomarkers of response to systemic treatment in Renal Cell Cancer. | 2 years
  Using data from RNA sequencing of tumour tissues, the outcome is to identify novel biomarkers of response.
Radiological identification of biomarkers of response to systemic treatment in Renal Cell Cancer. | 2 years
  Using data from MRI imaging by analysis of the tumour microenvironment and machine learning interrogation of output data, the outcome is to identify novel biomarkers of response.
Biological identification of biomarkers of response to systemic treatment in Renal Cell Cancer. | 2 years
  Using data from immunohistochemistry, the outcome is to identify novel biomarkers of response.
Biological identification of biomarkers of response to systemic treatment in Renal Cell Cancer. | 2 years
  Using data from immunofluorescence, the outcome is to identify novel biomarkers of response.
Biological identification of biomarkers of response to systemic treatment in Renal Cell Cancer. | 2 years
  Using data from CyTOF (mass cytometry), the outcome is to identify novel biomarkers of response.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Welsh, Principal Investigator — Cambridge University Hospitals

IPD SHARING:
Plan to Share IPD: Undecided